CLINICAL TRIAL: NCT07214571
Title: A Phase 2b, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Safety, Tolerability, and Efficacy of S-337395 in Symptomatic Nonhospitalized Adults With Respiratory Syncytial Virus Who Are at High Risk of Progression to Severe Disease
Brief Title: A Study of S-337395 in Symptomatic Nonhospitalized Adults With Respiratory Syncytial Virus (RSV) Who Are at High Risk of Progression to Severe Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2402T1432
Record Dates: First submitted 2025-10-08; First posted 2025-10-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory Syncytial Virus Infections; RSV infection; Viral infection; S-337395; Acute lower respiratory tract infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- S-337395 High Dose (Experimental): Participants will receive a high dose of S-337395 twice daily (BID) orally for up to 5 days.
  Interventions: Drug: S-337395
- S-337395 Low Dose (Experimental): Participants will receive a low dose of S-337395 BID orally for up to 5 days.
  Interventions: Drug: S-337395
- Placebo (Placebo Comparator): Participants will receive matching placebo BID orally for 5 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S-337395 — S-337395 will be administered per schedule specified in the arm description.
  Arms: S-337395 High Dose; S-337395 Low Dose
Drug: Placebo — Placebo matched to S-337395 will be administered per schedule specified in the arm description.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to investigate the antiviral effect of S-337395 compared with placebo among nonhospitalized adult participants with high-risk factors for progression to severe RSV infection starting intervention within 72 hours of RSV symptom onset.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants who have new onset or worsening (if present chronically) of at least 1 of the following signs and/or symptoms consistent with a viral acute respiratory infection within 72 hours prior to randomization: fever, nasal congestion, nasal discharge, sore throat, cough, sputum production, shortness of breath, or wheezing.
* Participants diagnosed with RSV infection preferably using a rapid polymerase chain reaction (PCR) or other molecular-based diagnostic assay.
* Has at least 1 of the following risk factors for severe RSV disease:

  1. ≥ 75 years of age;
  2. Chronic lung disease that is symptomatic and requiring chronic treatment; and
  3. Chronic cardiovascular disease that is symptomatic and requiring chronic treatment.
* With the exception of the RSV disease, medically stable on the basis of medical history, physical examination, vital signs, and 12-lead electrocardiogram (ECG) performed at screening.

Key Exclusion Criteria:

* Hospitalized or expected to be hospitalized within 24 hours of screening.
* Is considered by the investigator to be immunocompromised, due to an underlying medical condition or medical therapy, chemotherapy, radiation, stem cell or solid organ transplant.
* Has known allergies, hypersensitivity, or intolerance to S-337395 or to any of the excipients of the S-337395 or placebo formulation.
* Suspicion or known severe renal impairment.
* Any other medical or psychiatric condition making the participant unsuitable for the current study or interfering with the evaluation of response to the study intervention in the opinion of the investigator/subinvestigator.
* Has received a therapy intended to treat RSV infection within 14 days prior to screening.
* Is receiving chemotherapy or immunotherapy for malignancy.
* Has received RSV vaccination within 7 days prior to screening.
* Has had either confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) or influenza infection (test was positive) during the 28 days prior to screening.
* Has any other confirmed clinically relevant respiratory infection by any pathogen at, or within 28 days of screening.

Note: Other protocol-specified inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in RSV Ribonucleic Acid (RNA) Load by Quantitative Reverse Transcription Polymerase Chain Reaction (qRT-PCR) (Nasopharyngeal Swab) at Day 2 | Baseline, Day 2
Change From Baseline in RSV RNA Load by qRT-PCR (Nasopharyngeal Swab) at Day 4 | Baseline, Day 4
Change From Baseline in RSV RNA Load by qRT-PCR (Nasopharyngeal Swab) at Day 6 | Baseline, Day 6

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Day 1 up to Day 28
Change From Baseline in Severity of RSV Respiratory Symptom Score Based on the Respiratory Infection Intensity and Impact Questionnaire (RiiQ) Respiratory Symptom Subscale (RiiQ-RSS) | Baseline up to Day 6
Change From Baseline in Severity of RSV Systemic Symptoms Score Based on the RiiQ Systemic Symptom Subscale (RiiQ-SSS) | Baseline up to Day 6
Change From Baseline in Severity of RSV Total Symptoms Score Based on the Combined RiiQ RSS and RiiQ-SSS | Baseline up to Day 6
Time to First Resolution of All Respiratory RSV-related Symptoms Based on the RiiQ-RSS | Baseline up to Day 6
Time to Sustained (2 Consecutive Days) Resolution of All Respiratory RSV-related Symptoms Based on the RiiQ-RSS | Baseline up to Day 6
Time to First Resolution of All Systemic RSV-related Symptoms Based on the RiiQ-SSS | Baseline up to Day 6
Time to Sustained Resolution of All Systemic RSV-related Symptoms Based on the RiiQ-SSS | Baseline up to Day 6
Time to First Resolution of All Respiratory and Systemic RSV-related Symptoms Based on the Combined RiiQ RSS and RiiQ-SSS | Baseline up to Day 6
Time to Sustained Resolution of All Respiratory and Systemic RSV-related Symptoms Based on the Combined RiiQ RSS and RiiQ-SSS | Baseline up to Day 6
Time to First Resolution of Each Separate RSV-related Symptom Based on the RiiQ Symptom Subscale | Baseline up to Day 6
Time to Sustained Resolution of Each Separate RSV-related Symptom Based on the RiiQ Symptom Subscale | Baseline up to Day 6
Change From Baseline in RSV RNA Load | Baseline up to Day 6
Area Under the Curve (AUC) of Change From Baseline in RSV RNA Load | Baseline up to Day 6
Time to the First Negative RSV RNA Load by qRT-PCR | Baseline up to Day 6
Time to Sustained Negative RSV RNA Load by qRT-PCR | Baseline up to Day 6
Percentage of Participants With Negative RSV RNA Load by qRT-PCR | Baseline up to Day 6
Time to the First RSV RNA Load <Lower Limit of Quantitation (LLOQ) | Baseline up to Day 6
Time to Sustained RSV RNA Load <LLOQ | Baseline up to Day 6
Percentage of Participants With RSV RNA Load <LLOQ | Baseline up to Day 6
Change From Baseline in Infectious Titer | Baseline up to Day 6
AUC of Change From Baseline in Infectious Titer | Baseline up to Day 6
Time to the First Negative RSV Infectious Titer | Baseline up to Day 6
Time to Sustained Negative RSV Infectious Titer | Baseline up to Day 6
Percentage of Participants With Negative RSV Infectious Titer | Baseline up to Day 6
Time to the First RSV Infectious Titer <LLOQ | Baseline up to Day 6
Time to Sustained RSV Infectious Titer <LLOQ | Baseline up to Day 6
Percentage of Participants With RSV Infectious Titer <LLOQ | Baseline up to Day 6
Plasma Concentration of S-337395 After Repeated Oral Doses of S-337395 | Baseline up to Day 6
Plasma Concentration of S-337395 12 and 24 Hours After the First Dose and the Last Dose (C12 and C24) | 12 hours and 24 hours after first dose (Day 2) and last dose (Day 6)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (17):
  - Med Partnes, Inc - Elligo- PPDS, Toluca Lake, California
  - Doral Medical Research, Hialeah, Florida
  - Southern Clinical Research, Miami, Florida
  - Nuren Medical and Research Center, Miami, Florida
  - Continental Clinical Research, LLC, Miami, Florida
  - Dynamic Medical Research, LLC - Miami, Miami, Florida
  - Miami Clinical Research, LLP., Miami, Florida
  - Oceanic Research Group, LLC, North Miami Beach, Florida
  - CDC Research Institute, LLC, Port Saint Lucie, Florida
  - Cordova Research Insittute, Sweetwater, Florida
  - Better Life Clinical Research LLC, Tampa, Florida
  - Research Bay,Inc., Tampa, Florida
  - Santos Research Center - 5927 Webb Rd, Tampa, Florida
  - Covenant Pulmonary Criticial Care and Research Ins, East Point, Georgia
  - Clay Platte Family Medicine - CCT Research, Kansas City, Missouri
  - Prime Global Research, Inc., The Bronx, New York
  - Clinical Research Partners LLC, Richmond, Virginia
- Japan (26):
  - Kamezawa Clinic, Kasugai-Shi, Aiti
  - Doi Clinic, Chikushino-shi, Fukuoka
  - Irie Clinic, Fukuoka, Fukuoka
  - PS Clinic, Fukuoka-Shi Hakata-Ku, Fukuoka
  - Medical corporation Aimeikai Morizono internal medicine, Kitakyushu-Shi Yahatanishi-Ku, Fukuoka
  - Social Medical Corporation the Chiyukai foundation Shin Komonji Hospital, Kitakyushu-Shi, Fukuoka
  - Shizuka Clinic, Takasaki-shi, Gunma
  - Social medical corporation Keiwakai Nishioka Hospital, Sapporo-Shi Toyohira-Ku, Hokkaidô
  - Terada Internal Medicine and Respiratory Department, Himeji-shi, Hyôgo
  - Tsuchiura Beryl Clinic, Tsuchiura-Shi, Ibaraki
  - Gajyumaru Clinic Tsukuba, Tsukuba, Ibaraki
  - Shiwa Central Pediatrics, Shiwa-gun, Iwate
  - Medical corporation Kojinkai Takahashi Internal Medicine, Kawasaki-Shi, Kanagawa
  - Ebino Centro Clinic, Ebino, Miyazaki
  - Rinku General Medical Center, Izumisano, Osaka
  - Yamaichi Building Internal Medicine Clinic, Adachi-Ku, Tokyo
  - Medical Corporation Hosoda Clinic, Katsushika-ku, Tokyo
  - Medical Corporation Shirayurikai Swing Building Nozaki Clinic, Musashino, Tokyo
  - Noguchi Internal Medicine Clinic, Nakano-Ku, Tokyo
  - Sato Clinic, Shibuya-Ku, Tokyo
  - Mih Clinic Yoyogi, Shibuya-Ku, Tokyo
  - Medical corporation Hiroyukai Yotsuya Internal Medicine, Shinjuku-Ku, Tokyo
  - Yoshida Clinic, Suginami-ku, Tokyo
  - Sekino Hospital, Toshima-Ku, Tokyo
  - Kijima Kids Clinic, Higashiokitama-gun, Yamagata
  - Toda Internal Medicine and Neurology, Hyōgo